CLINICAL TRIAL: NCT02953704
Title: Prospective, Longitudinal, Non-Interventional Study of Disease Burden and Treatment of Patients With Low-Risk Myelofibrosis (MF) or High-Risk Essential Thrombocythemia (ET) or ET Patients Receiving ET-Directed Therapy
Brief Title: Myelofibrosis and Essential Thrombocythemia Observational Study (MOST)
Status: Completed | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB-MA-MF-401
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Myelofibrosis; essential thrombocythemia; clinical characteristics; disease burden; patient-reported outcomes
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myelofibrosis Cohort: Patients will be categorized as low-risk using Dynamic International Prognostic Scoring System (DIPSS) risk OR intermediate-1 risk by DIPSS by reason of age alone.
- Essential Thrombocythemia Cohort: Patients will be age ≥ 60 years OR have history of thromboembolic events OR currently receiving ET-directed therapy.

SUMMARY:
The purpose of this prospective, longitudinal, noninterventional study is to describe clinical characteristics, evolution of disease burden, and treatment patterns in patients with select subcategories of essential thrombocythemia (ET) or myelofibrosis (MF).

ELIGIBILITY:
Inclusion Criteria:

* MF cohort: Diagnosis of MF and low-risk using DIPSS risk categorization OR intermediate-1 risk by DIPSS by reason of age alone.
* ET cohort: Diagnosis of ET and age ≥ 60 years OR history of thromboembolic events OR currently receiving ET-directed therapy (eg, hydroxyurea, anagrelide, interferon, busulfan, ruxolitinib, etc).
* Willing and able to provide written informed consent.
* Willing and able to complete patient assessment questionnaires either alone or with minimal assistance from a caregiver and/or trained site personnel.
* Under the supervision of a physician for the current care of MF or ET.

Exclusion Criteria:

* Individuals who are participating in blinded investigational drug studies.
* Individuals who are participating in Incyte investigational/interventional drug trials (company- or investigator-sponsored studies) until they have completed the 30-day end of study visit.
* Life expectancy ≤ 6 months.
* Diagnosis of secondary acute myeloid leukemia, myelodysplastic syndrome, chronic myelogenous leukemia, or secondary thrombocytosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from up to 250 community and academic centers across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1469 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Description of the clinical characteristics and evolution of disease burden in essential thrombocythemia (ET) and myelofibrosis (MF) patients | Approximately every 6 months through end of study, up to approximately 36 months

SECONDARY OUTCOMES:
Description of patterns of treatment, therapies, and clinical management | Approximately every 3-6 months through end of study, up to at least 36 months
Description of disease progression over time | Approximately every 3-6 months through end of study, up to at least 36 months
Describe hematocrit, hemoglobin, white blood cell (WBC) count, and platelet counts over time | Approximately every 3-6 months through end of study, up to at least 36 months
Description of the comorbidities associated with disease and progression | Approximately every 3-6 months through end of study, up to at least 36 months
Description of changes in patient-reported symptoms and quality of life (QOL) | Approximately every 3-6 months through end of study, up to at least 36 months
Description of the rate and time to leukemic transformation | Approximately every 3-6 months through end of study, up to at least 36 months
Description of rate of all-cause mortality and aggregate causes of mortality | Approximately every 3-6 months through end of study, up to at least 36 months
Description of reasons for patient ineligibility based on Dynamic International Prognostic Scoring System (DIPSS) during screening (MF patients only) | At screening
Description of time to first disease-related intervention or first progression event during the period of observation (MF patients only) | Baseline to end of study, up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn M. Scherber, MD, MPH, Study Director — Incyte Corporation
Locations (116):
- United States (114):
  - Huntsville, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Berkeley, California
  - Highland, California
  - Long Beach, California
  - Oceanside, California
  - Palo Alto, California
  - Santa Rosa, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Fort Collins, Colorado
  - Middletown, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Columbus, Georgia
  - Marietta, Georgia
  - Thomasville, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Harvey, Illinois
  - Maywood, Illinois
  - Normal, Illinois
  - River Forest, Illinois
  - Skokie, Illinois
  - Anderson, Indiana
  - Avon, Indiana
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Ames, Iowa
  - Topeka, Kansas
  - Westwood, Kansas
  - Danville, Kentucky
  - Mount Sterling, Kentucky
  - Paducah, Kentucky
  - Alexandria, Louisiana
  - Covington, Louisiana
  - Marrero, Louisiana
  - Rockport, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Columbia, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Jackson, Minnesota
  - Lansing, Minnesota
  - Bolivar, Missouri
  - Cape Girardeau, Missouri
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Kalispell, Montana
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Brick, New Jersey
  - East Orange, New Jersey
  - Florham Park, New Jersey
  - Morristown, New Jersey
  - Paramus, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - East Setauket, New York
  - Elmira, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Boone, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Hendersonville, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Tualatin, Oregon
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Dunmore, Pennsylvania
  - Gettysburg, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Willow Grove, Pennsylvania
  - Lancaster, South Carolina
  - Spartanburg, South Carolina
  - Watertown, South Dakota
  - Jackson, Tennessee
  - Amarillo, Texas
  - Arlington, Texas
  - Beaumont, Texas
  - Bryan, Texas
  - Dallas, Texas
  - Houston, Texas
  - McAllen, Texas
  - McKinney, Texas
  - Mesquite, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Bristol, Virginia
  - Seattle, Washington
  - Yakima, Washington
  - Martinsburg, West Virginia
  - Milwaukee, Wisconsin
- Puerto Rico (2):
  - Bayamón
  - Ponce

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ritchie E, Al-Janadi A, Kessler C, Scherber R, Kalafut T, Ren H, Mesa R. Patient-reported outcomes of patients with myelofibrosis or essential thrombocythemia enrolled in the MOST study. Leuk Lymphoma. 2022 Dec;63(13):3138-3153. doi: 10.1080/10428194.2022.2113531. Epub 2022 Oct 7. PMID 36205505
- [Derived] Gerds AT, Lyons RM, Colucci P, Kalafut P, Paranagama D, Verstovsek S. Disease and Clinical Characteristics of Patients With a Clinical Diagnosis of Myelofibrosis Enrolled in the MOST Study. Clin Lymphoma Myeloma Leuk. 2022 Jul;22(7):e532-e540. doi: 10.1016/j.clml.2022.02.001. Epub 2022 Feb 8. PMID 35256316
- [Derived] Yacoub A, Lyons R, Verstovsek S, Shao R, Chu DT, Agrawal A, Sivaraman S, Colucci P, Paranagama D, Mascarenhas J. Disease and Clinical Characteristics of Patients With a Clinical Diagnosis of Essential Thrombocythemia Enrolled in the MOST Study. Clin Lymphoma Myeloma Leuk. 2021 Jul;21(7):461-469. doi: 10.1016/j.clml.2021.02.011. Epub 2021 Mar 1. PMID 33839074